CLINICAL TRIAL: NCT02816372
Title: Ultra Protective Ventilation Without Extracorporeal Circulation in Severe ARDS Patients (VT4ARDS)
Acronym: VT4ARDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL16_0082; 2016-A00503-48 (Other: ANSM)
Record Dates: First submitted 2016-06-24; First posted 2016-06-28 (Estimated); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tidal volume 4 ml/kg Predicted Body Weight (PBW) (Experimental)
  Interventions: Other: Tidal volume reduction to 4 ml/kg Predicted Body Weight (PBW)

INTERVENTIONS:
Other: Tidal volume reduction to 4 ml/kg Predicted Body Weight (PBW) — Tidal volume reduction to 4 ml/kg predicted body weight from inclusion to weaning PEEP trial

SUMMARY:
Despite the use of protective ventilation, neuromuscular blocking agent and prone position, ARDS mortality remains high (30%-50%) in observational studies, and pneumothorax rate in randomized controlled trial remains stable (10%). The driving pressure (the ratio of tidal volume over respiratory system compliance) has recently been strongly associated with ARDS mortality, suggesting that tidal volume reduction below 6ml/kg may offer mortality benefit. While extracorporeal CO2 removal technique are currently under investigation in association with tidal volume reduction

ELIGIBILITY:
Inclusion Criteria:

* invasive mechanical ventilation
* ARDS (Berlin definition) with PaO2/FiO2 ratio ≤ 150 mm Hg

Exclusion Criteria:

* Age below 18 year
* planned duration of invasive mechanical ventilation < 48 hours
* ARDS criteria present for more than 24 hours
* known or suspected intracranial hypertension
* known or suspected COPD
* chronic respiratory failure under long term oxygen or non-invasive ventilation
* pneumothorax or broncho-pleural fistula
* morbid obesity with body weight >1 kg/cm height
* sickle cell disease
* recent bone marrow transplantation, aplasia following chemotherapy
* burn injury on more than 30% of body surface
* severe hepatic cirrhosis (Child-Pugh score C)
* extracorporeal circulation life support
* pregnancy
* advance directives to withhold or withdraw life-sustaining treatment
* previous inclusion in present study
* patient under an exclusion period following inclusion in another biomedical study
* patient deprived of freedom, minor, subject under a legal protective measure
* lack of affiliation to social security as required by French regulation
* lack of written informed consent by patient or next of kin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-06-14 (Actual); Study Completion 2018-06-14 (Actual)

PRIMARY OUTCOMES:
Change in driving pressure | Baseline and 24 hours following inclusion
  Driving pressure is the difference between total respiratory system plateau pressure minus total positive end-expiratory pressure (PEEP)

SECONDARY OUTCOMES:
Rate of patients who achieved tidal volume reduction equal to 4 ml/kg predicted body weight | 48 hours following inclusion
Rate of pneumothorax | Day 90
Change in right ventricule/left ventricule area | Baseline and 24 hours following inclusion
  Echographic measurement of right ventricule/left ventricule

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon - Hôpital de la Croix Rousse, Lyon, France

REFERENCES:
- [Result] Richard JC, Marque S, Gros A, Muller M, Prat G, Beduneau G, Quenot JP, Dellamonica J, Tapponnier R, Soum E, Bitker L, Richecoeur J; REVA research network. Feasibility and safety of ultra-low tidal volume ventilation without extracorporeal circulation in moderately severe and severe ARDS patients. Intensive Care Med. 2019 Nov;45(11):1590-1598. doi: 10.1007/s00134-019-05776-x. Epub 2019 Sep 23. PMID 31549225